CLINICAL TRIAL: NCT06303362
Title: Effects of Elastic Band Excercises on Chest Expansion in Patients With Forward Head Posture
Brief Title: Effects of Elastic Band Excercises on Chest Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/014258 Sumbal Nawaz
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Forward Head Posture
Keywords: forward head posture; chest expansion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic band excercises (Experimental): Elastic band excercises and stretching is given to shoulder muscles (deep neck flexors, pectoralis major and minor, rhomboids and trapezius)
  Interventions: Other: Elastic band excercise
- strengthening with conventional physical therapy (Active Comparator): strengthening with conventional physicaltherapy is given to shoulder muscles (deep neck flexors, pectoralis major and minor, rhomboids and trapezius)
  Interventions: Other: strengthening with conventional physical therapy

INTERVENTIONS:
Other: Elastic band excercise — experimenatal group was given elastic band excercises along with stretching (pectoralis major, minor, trapezius, rhomboids and neck flexors) and conventional therapy. Sessions will be given 3 days in a week for a period of 4 weeks. The assessment was done at baseline, after 2 weeks and at the end of 4 weeks.
  Arms: Elastic band excercises
Other: strengthening with conventional physical therapy — control group was given strengthening excercises and stretching (pectoralis major, minor, trapezius, rhomboids (Sessions will be given 3 days in a week for a period of 4 weeks. The assessment was done at baseline, after 2 weeks and at the end of 4 weeks.
  Arms: strengthening with conventional physical therapy

SUMMARY:
• To determine the effects of Elastic Band Exercises on Chest Expansion, Forward Head Posture and disability

DETAILED DESCRIPTION:
According to literature review elastic band exercises have been proposed as an effective intervention to correct FHP. However, no previous study done to see the effect of elastic band exercises on chest expansion along with correction of FHP. Therefore, this study will show the effectiveness of elastic band exercises on chest expansion in patients with FHP.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Age group Between 18 to 30 years
3. Forward head posture measured through craniovertebral angle less than 50 degrees
4. Chest expansion measurement values at axillary level less than 5.1 cm
5. MMT of upper limb greater than 4

Exclusion Criteria:

1. Any cardiopulmonary pathology
2. Recent rib fracture
3. Participants with other upper limb musculoskeletal pathologies
4. Spinal or any associated chest surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Cloth tape measurement | 4 weeks
  The common tool in practice to measure chest expansion is non-elastic tape measurement technique. To measure Chest expansion there are three anatomical landmarks which are used to measure chest wall mobility. To measure upper chest, wall mobility landmark is axillary, to measure middle chest wall mobility landmark is 4th intercostal space and to measure lower chest wall mobility landmark is xiphoid process.According to general criteria its values are 1.4cm (poor), 3.1cm (moderate) and 5.1cm (good). Sessions will be given 3 days in a week for a period of 4 weeks. The assessment was done at baseline, after 2 weeks and at the end of 4 weeks
Neck Disability Index | 4 weeks
  The neck disability index questionnaire accesses pain and associated disability. It is a 10 items of self-reported questionnaire. Each question has 5 score with a total maximum score of 50 points. The patient is advised to select one option for each question that best reflects the intensity of pain and their discomfort.The assessment was done at baseline, after 2 weeks and at the end of 4 weeks
Craniovertebral angle | 4 weeks
  Two lateral photographs were taken to determine the craniovertebral angle (CVA) and to analyze these photographs a measuring instrument known as Web Plot Digitizer was used. Through this software craniovertebral angle(CVA) was measured. This mobile application assessing forward head posture(FHP) in the form of craniovertebral angle. The patient was instructed to stand in front of camera and picture was taken. One point was on C7 spinous process, one was on tragus of ear and other point is the intersection of a horizontal line passing through the C7 spinous process and then craniovertebral angle was formed.The assessment was done at baseline, after 2 weeks and at the end of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin G, Zhao X, Wang W, Wilkinson T. The relationship between forward head posture, postural control and gait: A systematic review. Gait Posture. 2022 Oct;98:316-329. doi: 10.1016/j.gaitpost.2022.10.008. Epub 2022 Oct 14. PMID 36274469
- [Background] Balthillaya GM, Parsekar SS, Gangavelli R, Prabhu N, Bhat SN, Rao BK. Effectiveness of posture-correction interventions for mechanical neck pain and posture among people with forward head posture: protocol for a systematic review. BMJ Open. 2022 Mar 9;12(3):e054691. doi: 10.1136/bmjopen-2021-054691. PMID 35264350